CLINICAL TRIAL: NCT00043459
Title: Study of T900607-Sodium in Previously Treated Patients With Non-Hodgkin's Lymphoma.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Tularik (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-607-007
Record Dates: First submitted 2002-08-08; First posted 2002-08-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-03

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

INTERVENTIONS:
Drug: intravenous T900607-sodium

SUMMARY:
The purpose of the study is to determine whether T900607-sodium is effective and safe in treating non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed diagnosis of non-Hodgkin's lymphoma (NHL)
* Subjects must have received prior chemotherapy for their NHL
* At least 18 years of age
* Bidimensionally measurable disease amenable to CT scanning. At least one lesion must be least 1 X 1 cm in size.
* Karnofsky performance status of at least 70%
* Estimated life expectancy of at least 12 weeks
* Females of childbearing potential must have a negative pregnancy test and agree to use an effective contraceptive
* Subject must be able to comply with study procedures and follow-up examinations.
* Signed written informed consent
* Lab Values (obtained ≤ 7 days prior to study enrollment):
* ANC at least 1.5x10e9/L,
* Platelet count at least 100x10e9/L,
* Hemoglobin at least 8.5 g/dL,
* Creatinine within 2 times upper limit of normal,
* AST and ALT within 3 times upper limit of normal,
* Bilirubin within 1.5 times upper limit of normal,
* Albumin great than 2.5 g/dL,

Exclusion Criteria

* Severe, concurrent disease, infection or co-morbidity that, in the judgment of the investigator, would make the subject inappropriate for enrollment
* NYHA Class III/IV cardiac disease, left ventricular ejection fraction (LVEF) of <50%, or acute anginal symptoms
* Patients who have received any investigational agent within 4 weeks of enrollment
* Patients who are pregnant or breast-feeding
* History of prior malignancy other than NHL within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* History of central nervous system metastases or carcinomatous meningitis
* Major surgery within 4 weeks of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2002-07; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Boyd, Study Chair — Tularik
Locations (5):
- United States (5):
  - Scripps Health Center, La Jolla, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Rush Medical Center, Chicago, Illinois
  - Weill Medical College of Cornell University, New York, New York